CLINICAL TRIAL: NCT04431219
Title: First in Human Study for the Assessment of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Multiple Ascending Intravenous Doses of LIS1 in Kidney Transplanted Patients
Brief Title: First in Human Study: LIS1, an Induction Treatment in Kidney Transplanted Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenothera SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XT-1901
Record Dates: First submitted 2020-05-28; First posted 2020-06-16 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Kidney Transplant
Keywords: immunosuppression; polyclonal IgG; allograft transplantation; induction treatment; acute graft rejection

STUDY DESIGN:
Intervention Model Description: This is a phase I/II interventional, uncontrolled, single center, open-label study with an adaptive design conducted in two cohorts: Ascending Dose (AD) cohort and Therapeutic Dose (TD) cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascending Dose Cohort (Experimental): The AD cohort will be first recruited and will include 5 patients: 1 patient per dose, sequentially recruited, the recruitment of the next dose level patient will be assessed by Data Safety Monitoring Board :
  * Patient 1: 0.6 mg/Kg/day
  * Patient 2: 1 mg/Kg/day
  * Patient 3: 3 mg/Kg/day
  * Patient 4: 6 mg/Kg/day
  * Patient 5: 8 mg/Kg/day
  Once the 5 AD patients complete LIS1 treatment, the sponsor and the DSMB will rule on the LIS1 dose to obtain an optimal CD3+ cells depletion, with a good safety profile and will determine the therapeutic dose.
  Interventions: Biological: LIS1
- Therapeutic Dose Cohort (Experimental): The TD cohort will be recruited once the therapeutic dose is defined. This cohort will be divided in 2 subgroups of respectively 2 and 3 patients sequentially recruited.
  DSMB will review the safety and efficacy profile of the first 2 patients (Subgroup1) and decide:
  * To continue at the same dose and recruit the next 3 patients of Subgroup 2
  * To recruit the next 3 patients with a lower dose, estimated from AD as bringing efficient depletion
  * To recruit the next patient with a higher dose (+2 mg/kg), if the depletion is not considered satisfactory and if the safety profile is considered acceptable
  * To end the trial if LIS1 toxicity is too important vs its efficacy in CD3+ depletion.
  If the decision to increase the dose after the first two TD patients is made, an additional DSMB review will be planned after patient 8. The DSMB will decide to maintain the dose for the last 2 patients or to get back to the previous dose
  Interventions: Biological: LIS1

INTERVENTIONS:
Biological: LIS1 — LIS1 is an induction treatment on top of maintenance immunosuppressive regimen. All patients from AD and TD cohort will receive the conventional immunosuppressive regimen: tacrolimus (0.2 mg/kg) / mycophenolic acid (MMF, 2x1000 mg) / prednisone (20 mg from day 2). This conventional treatment should be started and monitored for all patients independently of their participation in the clinical trial. Methylprednisolone 500 mg / 100 mL saline / 30 minutes will be administered before reperfusion during the surgery and on post operation day 1 just before LIS1 administration.

SUMMARY:
This first in human study aims at evaluating LIS1, a stabilized solution of purified anti-T lymphocytes polyclonal glyco-humanized swine IgG with immunosuppressive activity, in regards of safety, T cell depletion, and pharmacokinetics / pharmacodynamics in 10 kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be listed for kidney transplantation,
* AD cohort participants: First transplantation, Panel Reactive Antibody (PRA) < 20%, negative Donor Specific Antibody (DSA), no anti-HLA antibodies, Epstein-Barr Virus positive (EBV+) serology,
* TD cohort participants: First transplantation, 0-50 % PRA, negative DSA, negative flow cytometry crossmatch (FCXM) for any patients with anti-HLA antibodies on screening is mandatory, Epstein-Barr Virus positive (EBV+) serology
* Participants must weigh at least 50 kg and have a Body Mass Index (BMI) 18.0 ≤ BMI < 35.0 kg/m2,
* White Blood Cells > 3000/mm3, platelets > 75000/mm3,
* Female participants (WOCBP) must have a negative pregnancy test at screening and use a highly effective birth control until 90 days after the last administration of study drug,
* Non-vasectomized male subjects having a female partner of childbearing potential must agree to the use of a highly effective method of contraception until 90 days after the last administration of study drug,
* Participants must be capable of giving signed informed consent.

Exclusion Criteria:

* Patients with an active cancer or a history of kidney cancer,
* Patients who have previously been exposed to other anti-lymphocyte globulins,
* Patients with previous organ transplantation,
* Patients with a history of specific viral infection that would contraindicate depleting antibody therapy (Hepatitis B and C, HIV),
* Patients with a positive HIV and/or Hepatitis B and C tests
* Patients who have uncontrolled concomitant bacterial or viral infections (unresolved during screening), mycosis and/or parasitosis,
* Patients with a significant liver function impairment: enzyme (AST and/or ALT) values must not exceed 1.5 times upper limit of normal,
* Patients with positive testing for tuberculosis (using QuantiFERON-TB test), Patients with CMV D+/R- constellation at transplant,
* Patients with seronegative EBV prior to transplantation,
* Patients who have previously been exposed to antibodies of swine origin,
* Expanded Criteria Donor (ECD) defined as donor older than 60 years,
* Participants who have participated in another research study involving an investigational product in the previous 3 months,
* Patients with cardiovascular or severe respiratory comorbidities (severe chronic respiratory failure, severe pulmonary fibrosis, obesity-ventilation syndrome, severe idiopathic pulmonary arterial hypertension) not allowing general anesthesia,
* Patients with type 1 diabetes,
* Participants who are pregnant, breast feeding or planning pregnancy during the study,
* Participants who have any form of substance abuse (drug, alcohol…), any other health abnormalities (psychiatric disorders) or condition that according to the investigator's opinion might endanger patient during his/her participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Safety of the treatment with LIS1: Blood pressure | up to 3 months after the transplant
  Clinical safety parameters (1): Systolic and diastolic blood pressure (mm Hg).
Safety of the treatment with LIS1: Pulse rate | up to 3 months after the transplant
  Clinical safety parameters (2): Pulse rate (beats per minute [bpm]) .
Safety of the treatment with LIS1: Body temperature | up to 3 months after the transplant
  Clinical safety parameters (3): Body temperature (Celsius degrees).
Safety of the treatment with LIS1: Graft rejection | up to 3 months after the transplant
  Clinical safety parameters (4): Graft rejection (yes/no).
Safety of the treatment with LIS1: Infection | up to 3 months after the transplant
  Clinical safety parameters (5): Viral infections (namely Cytomegalovirus [CMV], BK virus) (yes/no).
Safety of the treatment with LIS1: Re-admission | up to 3 months after the transplant
  Clinical safety parameters (6): Re-admission after patient discharge (yes/no).
Safety of the treatment with LIS1: Hospitalization | up to 3 months after the transplant
  Clinical safety parameters (7): Prolonged stay in hospital for >4 weeks (days).
Safety of the treatment with LIS1: CRP | up to 3 months after the transplant
  Laboratory parameters (1): C-Reactive Protein (CRP, mg/L).
Safety of the treatment with LIS1: LDH | up to 3 months after the transplant
  Laboratory parameters (2): Lactate Dehydrogenase (LDH, µkat/L).
Safety of the treatment with LIS1: aPTT | up to 3 months after the transplant
  Laboratory parameters (3): activated Partial Thromboplastin Time (aPTT, seconds).
Safety of the treatment with LIS1: Complete Blood Count (CBC) | up to 3 months after the transplant
  Laboratory parameters (4): Platelets (10^9/L), white blood cells (10^9/L), absolute neutrophil count (10^9/L), absolute lymphocyte count (10^9/L), absolute monocyte count (10^9/L), absolute eosinophil count (10^9/L), absolute basophil count (10^9/L).
Pharmacodynamics (depletion of T lymphocytes) of LIS1 | up to 3 months after the transplant
  Absolute T lymphocyte counts (10^9/L).

SECONDARY OUTCOMES:
Pharmacokinetics of LIS1 (1): swine IgG | up to 3 months after the transplant
  Serum concentration of swine IgG
Pharmacodynamics of LIS1 (2): cytokines | up to 3 months after the transplant
  Cytokine concentration (IL6, TNFα) (ng/mL).
Biology of LIS1 (1): electrolytes plasma concentration | up to 3 months after the transplant
  Plasma biochemistry: electrolytes (Na+, K+, Cl-, Ca++, Mg++, bicarbonates plasma concentrations mmol/L)
Biology of LIS1 (2): urea and creatinine | up to 3 months after the transplant
  Plasma biochemistry: urea and creatinine plasma concentration (mmol/L)
Biology of LIS1 (3): total plasma proteins | up to 3 months after the transplant
  Plasma biochemistry: Total protein plasma concentration (g/L)
Biology of LIS1 (4): plasmatic proteins | up to 3 months after the transplant
  Plasma biochemistry: electrophoresis of plasmatic proteins (percentages of albumin, alpha-1-globulin, alpha-2-globulin, beta-globulin, gamma-globulin)
Immunogenicity of LIS1 | up to 3 months after the transplant
  Detection of antidrug antibodies in serum

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ondrej Viklicky, Principal Investigator — Institut klinické a experimentální medicíny, Praha 4, Czech Republic
Locations (1):
- Institut klinické a experimentální medicíny, Prague, Czechia

REFERENCES:
- [Derived] Viklicky O, Slatinska J, Janousek L, Rousse J, Royer PJ, Toutain PL, Cozzi E, Galli C, Evanno G, Duvaux O, Bach JM, Soulillou JP, Giral M, Vanhove B, Blancho G. First-in-human Study With LIS1, a Next-generation Porcine Low Immunogenicity Antilymphocyte Immunoglobulin in Kidney Transplantation. Transplantation. 2024 Jul 1;108(7):e139-e147. doi: 10.1097/TP.0000000000004967. Epub 2024 Feb 29. PMID 38421879